CLINICAL TRIAL: NCT03818490
Title: Bergamot Aromatherapy for Anxiety in a Medical Office Among Children With Autism Spectrum Disorder: A Randomized, Controlled Trial
Brief Title: Aromatherapy for Anxiety Among Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Principal Investigator, Jessie Hawkins, PhD, Research Director, Nutraceuticals Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-1200
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Anxiety; Autism Spectrum Disorder
Keywords: Aromatherapy; Essential Oils; Children
MeSH Terms: conditions — Anxiety Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bergamot Aromatherapy (Experimental): Patients in this group inhaled bergamot essential oil for 15 minutes at the start of their medical office visit.
  Interventions: Other: Bergamot Aromatherapy
- Control (No Intervention): Patients in this group did not experience an intervention.

INTERVENTIONS:
Other: Bergamot Aromatherapy — Patients in this group inhaled bergamot essential oil for 15 minutes.
  Arms: Bergamot Aromatherapy

SUMMARY:
This study evaluated the use of bergamot aromatherapy in the treatment of anxiety in a medical office setting among children who are diagnosed with an autism spectrum disorder. H

DETAILED DESCRIPTION:
Bergamot aromatherapy relieves anxiety in adult populations but has not been tested in a pediatric population with autism spectrum disorder. Because autism spectrum disorders often include hypersensitivity to sensory experiences, the use of essential oils in this population should be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Between 6-11 years of age
* Diagnosed with an autism spectrum disorder

Exclusion Criteria:

* none

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline State Trait Anxiety Inventory for Children | baseline and after the 15 minute intervention
  Self reported anxiety survey measuring state anxiety in children through 20 questions with a score ranging from 0-60 with higher scores representing higher anxiety.
Change from baseline in Blood Pressure | baseline and after the 15 minute intervention
  Routine blood pressure measurement
Change from baseline in Heart Rate | baseline and after the 15 minute intervention
  Routine heart rate measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Franklin Institute of Wellness, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No